CLINICAL TRIAL: NCT06972810
Title: A Controlled Human Infection Study of a Recombinant H3N2 (A/Texas/71/2017, Clade 3C3a) Influenza Virus in Healthy Adults in Australia
Brief Title: Human Infection Study of H3N2 Influenza in Healthy Adults
Acronym: FluCHIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); WHO Collaborating Centre for Reference and Research on Influenza (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 27338
Record Dates: First submitted 2025-04-27; First posted 2025-05-15 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Influenza
Keywords: Influenza virus type A (H3N2); Challenge
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Influenza Challenge Model with Influenza A H3N2 virus strain (Experimental)
  Interventions: Other: A/Texas/71/2017, clade 3C3a H3N2 influenza virus

INTERVENTIONS:
Other: A/Texas/71/2017, clade 3C3a H3N2 influenza virus — The intervention product is a live challenge virus that is manufactured in the USA under Good Manufacturing Practice (GMP). The challenge will be administered intranasally using a sprayer device. Participants will be admitted into an inpatient facility prior to the administration of the flu virus. Following inoculation, they will be quarantined for a minimum of 8 days prior to discharge. Participants will receive supportive care and PCR positive participants will receive an effective antiviral medication. Participants will be followed for a total of 6 months.
  Other Names: A/Texas/71/2017, clade 3C3a H3N2

SUMMARY:
This study will examine how the immune system responds to a flu virus (H3N2) during and after infection in health adults aged between 18 and 50 while in an inpatient facility.

The study uses a specific flu virus called the H3N2 influenza challenge virus, that was produced specifically for use in clinical research in controlled conditions. From a previous study, mild to moderate symptoms are expected.

This is the first time that a flu challenge study has been undertaken in Australia.

DETAILED DESCRIPTION:
Influenza A and B viruses cause seasonal outbreaks that affect 2-10% of people in developed countries annually and contribute to up to 650,000 global deaths, according to the WHO. Transmission occurs via respiratory droplets, with most healthy adults recovering within a week. However, severe illness can occur in high-risk groups such as young children, the elderly, pregnant women, and individuals with comorbidities.

The self-limiting nature of influenza in healthy adults lends itself to controlled human infection models (CHIM) which offer key advantages for influenza research, including precise control over the virus strain, timing of infection, and the ability to collect well-timed pre- and post-infection samples.

Influenza challenge studies have provided key insights into host immune responses and supported the development of vaccines and antivirals.

This first-in-Australia influenza challenge study aims to evaluate the safety and infectivity of recombinant H3N2 (A/Texas/71/2017, clade 3C3a) in a serosusceptible cohort. The study will also explore early host-virus interactions using advanced immunological techniques, alongside viral shedding into the air through environmental sampling, the kinetics of viral transmission and microbiome changes.

ELIGIBILITY:
Inclusion Criteria:

1. General good health, without significant medical conditions that would interfere with participant safety, as defined by medical history, physical examination, screening laboratory tests, and ECG at a screening evaluation.
2. Susceptible to the challenge virus as determined by a baseline serum HAI and NAI antibody titer to the RG-A/Texas/71/2017 (H3N2; clade 3c3a) virus of 1:40 or less.
3. Able to understand and comply with planned study procedures and available for the duration of the trial.
4. Willing to participate in the study and adhere to all trial requirements, including providing written consent to remain at the trial site for at least seven days after administration of the challenge virus. This willingness must be demonstrated by signing the informed consent document.
5. Willing to allow the investigators to discuss the participant's medical history with their General Practitioner or any relevant health professional.
6. Willing to refrain from donating blood for the duration of the study period.
7. Willing to refrain from smoking and illicit drug use during the quarantine period.
8. Women of childbearing potential (WOCBP)* are required to practice a highly effective form of contraception during the course of the study. Acceptable forms of contraception for female participants include:

   1. Established use of oral, injected or implanted hormonal methods of contraception (established for a minimum of 4 weeks prior to first inpatient quarantine).
   2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).

      * Male sterilization, if the vasectomized partner is the sole partner for the participant and appropriate post vasectomy documentation of sterilization success is available.
   3. Same sex intercourse only.
   4. True abstinence from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the participant (Periodic abstinence and withdrawal are not acceptable methods of contraception). Careful history and documentation regarding the reliability of this method must be recorded.

Exclusion Criteria:

1. History of clinically significant or currently active neurological, cardiac, respiratory, hepatic, rheumatological, autoimmune, or renal disease. Specifically:

   1. History of chronic obstructive pulmonary disease, pulmonary hypertension, or chronic lung condition of any etiology;
   2. Current diagnosis of asthma or reactive airway disease (e.g., to viral infections) within the past 2 years;
   3. History of thromboembolic, cardiovascular or cerebrovascular disease;
   4. Current diabetes mellitus (Type I or Type II);
   5. Any history of malignancy except for non-recurrent basal cell carcinoma;
   6. History or evidence of clinically significant autoimmune disease or known immunodeficiency of any cause (including HIV);
   7. History of a surgical splenectomy;
   8. History of severe psychiatric illness at any time (e.g., psychiatric illness that resulted in inpatient admission, psychosis, suicide attempt) or current significant active symptoms of anxiety and/or depression; i. Participants with history of anxiety-related symptoms of any severity within the last 2 years if the Generalized Anxiety Disorder-7 score is ≥5 ii. Participants with a history of depression of any severity within the last 2 years if the Patient Health Questionnaire-9 score is ≥4
   9. Bleeding disorder (e.g., factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following injections or venepuncture; OR
   10. Other conditions that, in the opinion of the Investigator, could interfere with a participant completing the study and necessary investigations.
2. Any clinical laboratory test parameters ≥ 1.5x upper limit of normal (ULN) unless deemed by the investigator to have no clinical significance.
3. Body Mass Index (BMI) of less than 18.5 or greater than 32.
4. Behavioral or cognitive impairment that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol.
5. The use of alcohol or psychoactive drugs/controlled substances in the past 12 months that:

   1. Has had a functional impact on the participant's life;
   2. Has resulted in or been a medical condition that required treatment; OR
   3. Could constitute abuse or misuse
6. Current use of illicit substance use, defined as a negative urine drug screen at screening and at admission (cannabis (THC), amphetamine, barbiturates, benzodiazepines, cocaine, ecstasy, methamphetamine, methadone, opiates, Phencyclidine (PCP)).
7. History of anaphylaxis.
8. Allergy to both Oseltamivir and Baloxavir.
9. Known allergy to two or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
10. Personal or family history a severe response to a viral infection including but not limited to:

    1. Guillain-Barré Syndrome;
    2. Clinically significant post-viral fatigue or other post-viral long-term sequalae.
11. Previous hospitalization with influenza or related complications.
12. Use of corticosteroids (including nasal sprays/inhaled preparations but excluding other topical preparations) or immunosuppressive drugs within 30 days prior to challenge.
13. Receipt of a live vaccine within 4 weeks or other vaccine within 2 weeks prior to enrollment.
14. Receipt of any investigational drug or vaccine within 3 months or 5.5 half-lives (whichever is greater).
15. Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to challenge.
16. Smoking or vaping:

    1. Current smoker defined as anyone who has smoked a nicotine product (including any vaping) at anytime in the month prior to enrollment; OR
    2. Significant past history of smoking (defined as ≥ 20 year pack history and ceased smoking <10 years ago).
17. Participants who share a household with someone at higher risk for influenza-related complications, including:

    1. Persons ≥65 years of age or <5 years of age;
    2. Persons with chronic pulmonary disease (e.g., asthma), chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, ischemic heart disease), metabolic disease (e.g., diabetes mellitus, renal dysfunction, haemoglobinopathies), immunosuppression, neurological and neurodevelopmental conditions,
    3. Children and teenagers who are receiving long-term aspirin therapy, OR
    4. Women who are pregnant or who are trying to become pregnant.
18. Infection with human immunodeficiency virus-1 (HIV-1), hepatitis C virus (HCV), or hepatitis B (HBV)
19. Clinically significant abnormalities on ECG (as determined by the study investigator).
20. Concurrent enrollment (or planned at anytime over the course of this trial) in a study which uses an investigational product or collects participant's blood.
21. Acute medical condition which is either undiagnosed/still being investigated at time of challenge, OR requiring new or adjustment of prescription medication use in the 30 days prior to challenge.
22. Any neurologic abnormality impairing the gag reflex or contributing to aspiration.
23. Significant abnormality altering the anatomy of the nose/nasopharynx or clinically significant nasal deviation or any other clinically significant nasal pathology.
24. Recent history (180 days prior to challenge) of nasal/sinus surgery or epistaxis requiring a medical procedure to control it (e.g., cauterisation, packing, the use of topical vasoconstrictors).
25. Current sinusitis.
26. Venous access deemed inadequate for the phlebotomy demands of the study.
27. Confirmed infection with influenza virus (on PCR) within the past 6 months prior to enrollment.
28. Receipt of a seasonal influenza vaccine in the past 6 months prior to enrollment or planned receipt in the first 2 months of the study.
29. Any condition or finding, to include medical and psychiatric conditions, that in the opinion of the Investigator, might interfere with the safety of the participant, affect the participant's ability to participate in the trial and/or interfere with the collection or interpretation of the study objectives.
30. Participants who are excluded from the study because they have been discovered during screening procedures to be suffering from a previously undiagnosed condition thought to require further medical attention will, with their consent, be referred appropriately to their GP or a specialist.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who become infected with the virus | Day 1 to Day 7 post challenge
  Confirmation of the challenge dose of virus to achieve a symptomatic influenza attack rate (AR) of 78% defined as:
  Percentage of participants with detectable shedding in nasopharyngeal (NP) swab(s) identified on RT-PCR over any 2 days between days 1-7 post challenge.
  AND Symptom score that meets the clinical case definition for symptomatic infection (modified Jackson score ≥ 6).
Safety of the H3N2 challenge model | Day 0 to 6 months post challenge
  Frequency and severity of adverse events (AEs) events, either self-reported, or observations, during inpatient confinement and at clinic visits throughout the study period.

SECONDARY OUTCOMES:
Detection of asymptomatic infection | Day 1 to 7 post challenge
  Percentage of participants who have detectable viral shedding in nasopharyngeal swabs by RT-PCR on any 2 days between days 1-7 post challenge AND who record a modified Jackson score < 6
Percentage of participants who develop influenza antibodies | Day 0 - 14 post challenge
  Percentage of participants who develop serological evidence of infection defined as a ≥ 4-fold rise in influenza-specific serum antibody

OTHER OUTCOMES:
Investigate associations between virus shedding, symptoms and immune responses of participant post virus inoculation | Day -2 (baseline) to Day 56
  Measure changes in peripheral blood H3N2-specific antibody levels, antigen-specific B cell frequencies, B and T cell receptor gene usage and expression, circulating cytokines and metabolites, and determine participant HLA genotype
Investigate associations between virus shedding and immune response kinetics and changes in the microbiome | Day -2 (baseline) to Day 56
  Measure any changes of the microbiome in the respiratory mucosa and/or stool pre- and post-infection
Determine whether influenza virus is shed into the air following challenge infection | Day 2 to Day 6 post challenge
  Air samples from participants post inoculation will be collected and assayed to determine whether infectious influenza virus or viral nucleic acid is exhaled.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Gail Cross, MBSS (BSc), FRACP, Principal Investigator — University of Melbourne
Locations (1):
- Doherty Clinical Trials, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided